CLINICAL TRIAL: NCT01219712
Title: Preoperative Optimization of the High-Risk Patient Undergoing Hip Fracture Surgery
Brief Title: Optimization Study of Cardiac Risk Patients With Hip Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Linkoeping (Other)
Collaborators: Region Örebro County (Other); Ryhov County Hospital (Other)
Responsible Party: Christina Eintrei, Department of Medical and Health Sciences, Division of drug research & anesthesiology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Hip-Op 101a
Record Dates: First submitted 2010-09-09; First posted 2010-10-13 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-09

CONDITIONS: Left Ventricular Dysfunction; Femoral Fracture
Keywords: NT-proBNP; non-cardiac surgery; left ventricular dysfunction; cardiac complications
MeSH Terms: conditions — Ventricular Dysfunction, Left; Femoral Fractures | interventions — Colloids; Dobutamine; Simendan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Preoperative Optimization (Active Comparator): Patients with proximal femur fracture who are > 65 yrs old and have an increased NT-proBNP would be randomized to either Standard Management or Optimized Management.
  The main aim of optimization is to achieve a normal oxygen delivery to the tissues preoperatively.
  * Hb would be optimized to > 90 g/l
  * SaO2 > 96%
  * Stroke volume index (SVI) > 30
  * Heart rate should ideally be < 80
  Stroke volume index (SVI) > 30 is achieved by repeated volume substitution in the form of 100-200 ml colloid. If, despite bolus doses of colloids, the SVI is < 30, one would have to use ionotropic drugs e.g. dobutamine or levosimendan, in order to achieve this goal.
  Interventions: Procedure: Colloids, dobutamin, levosimendan
- Standard treatment (No Intervention): Patients who are randomized to this group would be managed according to existing routines within the hospital. Consequently, these patients would be transferred to the Orthopaedic ward after initial management in the Emergency Department, including fluid therapy, oxygen and pain management. Since these patients have a significantly high NT-proBNP, a Cardiologist would be consulted and a decision for optimization taken together with the attending Anaesthesiologist and Orthopaedic Surgeon prior to surgery.
  Interventions: Procedure: Colloids, dobutamin, levosimendan

INTERVENTIONS:
Procedure: Colloids, dobutamin, levosimendan — : The main aim of goal-directed therapy is to achieve a normal oxygen delivery to the tissues i.e. DO2 500-600ml/min/m2.
  * Hb would be optimized to > 90 g/l
  * SaO2 > 96%
  * Stroke volume index (SVI) > 30
  * Heart rate should ideally be < 80
  Stroke volume index (SVI) > 30 is achieved by repeated volume substitution in the form of 100-200 ml colloid. If, despite bolus doses of colloids, the SVI is < 30, one would have to use ionotropic drugs e.g. dobutamine or levosimendan, in order to achieve this goal
  Other Names: Optimization; Hip fracture; Left ventricular dysfunction; Cardiac complication

SUMMARY:
Elderly patients undergoing surgery for proximal hip fracture have a high risk of morbidity and mortality (M&M) postoperatively. Several studies including some from the investigators department have shown that there is a high risk of cardiovascular complications in this group of patients and 3-month mortality is 15-20%. One of the causes of this high M&M is the high incidence of cardiac failure associated with an increased NT-proBNP in this group of patients. The aim of the present study is to evaluate whether optimization of preoperative cardiac function can reduce cardiac M&M postoperatively. Following verbal consent, patients with an increased NT-proBNP would be randomized to goal-directed preoperative optimization or standard management according to current hospital routines. Following optimization, the patients would be transferred to the operating rooms and subsequent management including perioperative patient management would be left to the discretion of a specialist anesthesiologist who is directly involved in patient care. Postoperatively, Troponin T and NT-proBNP would be measured in all patients according to the study protocol. In addition, major adverse cardiac events would be documented and follow-up would be done by after 30 days and 3 months postoperatively.

DETAILED DESCRIPTION:
This is a prospective, open, randomized, multi-center study. Primary screening of patients would take place in the Emergency room or Orthopedic ward according to the inclusion and exclusion criteria (see below). All patients (>= 65 yr) with a proximal hip fracture would be required to provide either written or verbal informed consent prior to being included in the study. Subsequently, NT-proBNP would be taken and if this is above the recommended levels suggesting cardiac failure (> 900 ng/l in patients 65-75 yrs old, and >1800 ng/l in patients > 75 yrs), the patients may be included into the study. Included patients would then be randomized into two groups: Standard management according to existing hospital routines and Optimized Management Patients with a normal NT-proBNP would be listed but would not be included in the study. Patients with proximal femur fracture who are > 65 yrs old and have an increased NT-proBNP and who have given informed consent would be randomized to either Standard Management or Optimized Management. The former group would be managed according to the hospital routines and cared for by a Specialist Anaesthesiologist and Orthopaedic surgeon preoperatively.

Group O= Optimization Patients who are randomized to the Optimization group would be transferred to a Holding Area, which is close to the Operating Rooms 4-6 hours prior to planned surgery. The main aim of optimization is to achieve a normal oxygen delivery to the tissues preoperatively i.e. DO2: 500-600ml/min/m2. Optimized management means that patients first have an Echocardiography to evaluate myocardial function. Subsequently, an arterial line is inserted and optimization achieved by using this arterial line connected to a Flo-track system (Vigileo, Edwards). The system uses pulse wave analysis to assess several parameters including: stroke volume index (SVI), cardiac index (CI), systemic vascular resistance index (SVRI), as well as oxygen delivery (DO2).The main aim of goal-directed therapy is to achieve a normal oxygen delivery to the tissues i.e. DO2 500-600ml/min/m2.• Hb would be optimized to > 90 g/l

* SaO2 > 96%
* Stroke volume index (SVI) > 30
* Heart rate should ideally be < 80

Stroke volume index (SVI) > 30 is achieved by repeated volume substitution in the form of 100-200 ml colloid. If, despite bolus doses of colloids, the SVI is < 30, one would have to use ionotropic drugs e.g. dobutamine or levosimendan, in order to achieve this goa

The study would be done in three hospitals: University Hospital, Linköping, University Hospital, Örebro and Jönköping Hospital. A total of 200 patients (100 in each group) would be included. It is expected that the study would be ongoing during a period of two years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients > 65 yrs
2. Proximal femur fracture where the patient is planned to be operated during the day (Monday-Friday).
3. NT-proBNP > 900 ng/l in patients 65-75 yrs old, and >1800 ng/l in patients > 75 yrs.
4. Informed consent provided by the patient.

All of the above criteria must be fulfilled before the patient can be included in the study.

Exclusion Criteria:

1. Informed consent cannot be provided
2. Mental or verbal difficulty in understanding or expressing willingness to participate in the study.
3. Instable angina pectoris.
4. Ongoing myocardial infarct or ischemia
5. Circulatory shock
6. Decompensated cardiac failure or pulmonary oedema
7. Pathologic femur fracture
8. Chronic haemodialysis
9. Cardiac valve incompetence that has haemodynamic consequences

Any one of the above is a criterion for exclusion.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Major cardiac complications | during hospital stay (approximately 10 days)
  myocardial injury (Troponin T ≥ 0.04 μg/l and/or myocardial infarct or death from cardiac complications or therapy-requiring cardiac failure)

SECONDARY OUTCOMES:
Mortality | 30 days
  all cause
Mortality | 3 months
  All cause
Length of hospital stay | 7-14 days

CONTACTS AND LOCATIONS:
Overall Officials: Christina Eintrei, Professon, Study Director — Department of Medical & Health Sciences Division of Drug Research/Anaesthesiology
Locations (3):
- Sweden (3):
  - Department of Anaesthesia & Intensive Care, Jönköping
  - Department of Anaesthesia & Intensive Care, University Hospital, Linköping
  - Department of Anaesthesia & Intensive Care, University Hospital, Örebro